CLINICAL TRIAL: NCT06551298
Title: Multi Center Clinical Study on the Lipid-lowering Efficacy and Safety of Menggongzi Tibetan Tea Special Drink
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chunjian Li, Director of Cardiology, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 032
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Hyperlipidemias
Keywords: Hyperlipidemias; Tibetan tea; Atorvastatin
MeSH Terms: conditions — Hyperlipidemias | interventions — Atorvastatin; Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental group (Experimental): Menggongzi Tibetan Tea Special Drink (50ml/time, taken after breakfast and lunch)+Low fat diet
  Interventions: Other: Menggongzi Tibetan Tea Special Drink
- Positive control group (Active Comparator): Atorvastatin Calcium Tablets (20mg, qn)+Low fat diet
  Interventions: Drug: Atorvastatin Calcium 20Mg Tab
- Negative control group (Other): Low fat diet
  Interventions: Other: Low fat diet

INTERVENTIONS:
Other: Menggongzi Tibetan Tea Special Drink — Menggongzi Tibetan Tea Special Drink (50ml/time, taken after breakfast and lunch)+Low fat diet
  Arms: Experimental group
Drug: Atorvastatin Calcium 20Mg Tab — Atorvastatin Calcium Tablets (20mg, qn)+Low Fat Diet
  Arms: Positive control group
Other: Low fat diet — Low fat diet
  Arms: Negative control group

SUMMARY:
About 179 million people die from cardiovascular disease each year, accounting for approximately 31% of global deaths. It is expected that this number will exceed 236 million by 2030, and the economic burden caused by this disease is increasing year by year.At present, the number of people suffering from cardiovascular diseases in China is as high as 330 million, and the mortality rate accounts for more than 40% of the total deaths caused by diseases, and is in a continuous upward trend.Long term dyslipidemia will increase the incidence rate and mortality of atherosclerotic diseases.Tibetan tea contains catechins, caffeine, amino acids, vitamins, and various mineral components, which have significant effects in reducing cholesterol, improving carbohydrate metabolism, lowering blood sugar, losing weight, softening human blood vessels, and other aspects.At present, there are no research reports on the lipid-lowering effect of Mongolian Gongzi Tibetan Tea Special Drink, and most studies on the lipid-lowering effect of Tibetan Tea are animal experiments or clinical observational studies. Therefore, this study intends to use a randomized controlled trial to explore the lipid-lowering efficacy and safety of Mongolian Gongzi Tibetan Tea Special Drink in patients with hyperlipidemia.

DETAILED DESCRIPTION:
Every year, approximately 179 million people die from cardiovascular diseases, accounting for about 31% of global deaths. This number is expected to exceed 236 million by 2030, and the economic burden of these diseases is increasing year by year. Currently, in China, there are up to 330 million people suffering from cardiovascular diseases, with the mortality rate exceeding 40% of disease-related deaths and continuing to rise. Chronic dyslipidemia increases the incidence and mortality of atherosclerotic cardiovascular disease (ASCVD). Hyperlipidemia refers to elevated levels of one or more lipids in the plasma due to abnormal lipid metabolism or transport, leading to deposition in the vascular endothelium and causing damage to the body. This condition manifests as hypercholesterolemia, hypertriglyceridemia, or low high-density lipoprotein cholesterol. Additionally, this disease is closely related to the onset of stroke, diabetes, hypertension, fatty liver, and other conditions. In recent years, the incidence of hyperlipidemia has significantly increased due to changes in lifestyle, especially dietary habits. The atherosclerotic cardiovascular diseases caused by hyperlipidemia are often characterized by high incidence, severe harm, and rapid disease progression. Hyperlipidemia is becoming an invisible killer of human health.

Statins are the most recommended medication for ASCVD due to their significant effect in lowering low-density lipoprotein cholesterol, with strong evidence supporting their use. However, the side effects of statins have not been fully resolved. Among patients receiving statin treatment, 10%-29% may experience statin-related muscle symptoms, such as cramps, myalgia, weakness, immune-mediated necrotizing myopathy, and more rarely, rhabdomyolysis. Medium-intensity statins may increase the risk of type 2 diabetes by approximately 11%, while high-intensity statins might increase the risk by 20% or more. Early clinical trials of statins showed that up to 2% of patients experienced elevated transaminases, and the impact on renal function remains controversial. Additionally, statin-related adverse events include cataracts, gastrointestinal issues, effects on the genitourinary system, gynecomastia, and reproductive issues. Balancing the benefits and risks of statin therapy is a crucial challenge for all cardiovascular doctors.

Tea is one of the world's three major non-alcoholic beverages and has been used both as a food and medicine for over 5000 years. Yaan Tibetan tea is a local specialty black tea, named after its primary production in Yaan, Sichuan Province, and historically popular in Tibetan areas such as Tibet and Qinghai. Tibetan tea contains catechins, caffeine, amino acids, vitamins, and various minerals, particularly rich in tea pigments, tea polysaccharides, and tea saponins. Besides the general benefits of tea such as anti-cancer, anti-aging, antioxidant, anti-bacterial, and anti-radiation effects, it has significant effects on lipid reduction, improving carbohydrate metabolism, lowering blood sugar, weight loss, and softening blood vessels. Meng Gongzi Tibetan Tea Special Drink is made from Tibetan tea, using modern green separation and purification technology to extract and concentrate key functional components like tea polysaccharides and tea pigments. It adds sorbitol, which is indigestible and harmless to the human body, to enhance palatability and is produced using instant sterilization and hot filling technology without preservatives, strictly according to GB/T21733 standards, resulting in a convenient drink with high tea pigment and polysaccharide content.

Currently, there is no research report on Meng Gongzi Tibetan Tea Special Drink, and studies on the lipid-lowering effects of Tibetan tea are mostly animal experiments or observational studies. Therefore, this study aims to use a randomized controlled trial to explore the lipid-lowering efficacy and safety of Meng Gongzi Tibetan Tea Special Drink for patients with hyperlipidemia.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria for hyperlipidemia: total cholesterol (TC) ≥ 6.20mmol/L, triglycerides (TG) ≥ 2.30 mmol/L. If one of the above blood lipid indicators is abnormal, it can be included in this study;
2. Age ≥ 18 years old, gender not limited;
3. The patient is willing to follow the research protocol and sign an informed consent form.

Exclusion Criteria:

1. Atherosclerotic cardiovascular disease (ASCVD) patients;
2. Diabetes patients;
3. Severe hypercholesterolemia (TC>8 mmol/L or LDL-C ≥ 4.9 mmol/L) or severe hypertriglyceridemia (TG ≥ 5.6 mmol/L);
4. Secondary hyperlipidemia;
5. Individuals with a family history of primary hypercholesterolemia;
6. Active liver disease or unexplained persistent elevation of serum transaminases (aspartate aminotransferase (AST) or alanine aminotransferase (ALT)>2-fold upper limit of normal (ULN));
7. The estimated glomerular filtration rate (eGFR) is less than 30 mL/min/1.73m2;
8. Creatine kinase (CK)>3 times ULN;
9. Individuals who have used any lipid-lowering drugs within the past month; 10）Individuals allergic to Tibetan tea and atorvastatin calcium;

11) Individuals with combined mental illnesses or malignant tumors; 12) Pregnant and lactating women; 13) Researchers consider patients who are not suitable for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-08-08 (Estimated); Study Completion 2025-08-08 (Estimated)

PRIMARY OUTCOMES:
TC | 4 weeks
  Comparison of TC levels between Tibetan tea and a simple low-fat diet compared to baseline
TG | 4 weeks
  Comparison of TG levels between Tibetan tea and atorvastatin compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139
- [Background] Zenych A, Fournier L, Chauvierre C. Nanomedicine progress in thrombolytic therapy. Biomaterials. 2020 Nov;258:120297. doi: 10.1016/j.biomaterials.2020.120297. Epub 2020 Aug 6. PMID 32818824
- [Background] Li Z, Lin L, Wu H, Yan L, Wang H, Yang H, Li H. Global, Regional, and National Death, and Disability-Adjusted Life-Years (DALYs) for Cardiovascular Disease in 2017 and Trends and Risk Analysis From 1990 to 2017 Using the Global Burden of Disease Study and Implications for Prevention. Front Public Health. 2021 Oct 29;9:559751. doi: 10.3389/fpubh.2021.559751. eCollection 2021. PMID 34778156
- [Background] writing committee of the report on cardiovascular health and diseases in china. Report on Cardiovascular Health and Diseases in China 2021: An Updated Summary. Biomed Environ Sci. 2022 Jul 20;35(7):573-603. doi: 10.3967/bes2022.079. PMID 35945174
- [Background] Adhyaru BB, Jacobson TA. Safety and efficacy of statin therapy. Nat Rev Cardiol. 2018 Dec;15(12):757-769. doi: 10.1038/s41569-018-0098-5. PMID 30375494
- [Background] Colantonio LD, Huang L, Monda KL, Bittner V, Serban MC, Taylor B, Brown TM, Glasser SP, Muntner P, Rosenson RS. Adherence to High-Intensity Statins Following a Myocardial Infarction Hospitalization Among Medicare Beneficiaries. JAMA Cardiol. 2017 Aug 1;2(8):890-895. doi: 10.1001/jamacardio.2017.0911. PMID 28423147
- [Background] Sattar N. Statins and diabetes: What are the connections? Best Pract Res Clin Endocrinol Metab. 2023 May;37(3):101749. doi: 10.1016/j.beem.2023.101749. Epub 2023 Feb 15. PMID 36858834
- [Background] Khatiwada N, Hong Z. Potential Benefits and Risks Associated with the Use of Statins. Pharmaceutics. 2024 Feb 1;16(2):214. doi: 10.3390/pharmaceutics16020214. PMID 38399268
- [Background] Ward NC, Watts GF, Eckel RH. Statin Toxicity. Circ Res. 2019 Jan 18;124(2):328-350. doi: 10.1161/CIRCRESAHA.118.312782. PMID 30653440
- [Background] Bakker-Arkema RG, Davidson MH, Goldstein RJ, Davignon J, Isaacsohn JL, Weiss SR, Keilson LM, Brown WV, Miller VT, Shurzinske LJ, Black DM. Efficacy and safety of a new HMG-CoA reductase inhibitor, atorvastatin, in patients with hypertriglyceridemia. JAMA. 1996 Jan 10;275(2):128-33. PMID 8531308
- [Background] Ginsberg HN, Packard CJ, Chapman MJ, Boren J, Aguilar-Salinas CA, Averna M, Ference BA, Gaudet D, Hegele RA, Kersten S, Lewis GF, Lichtenstein AH, Moulin P, Nordestgaard BG, Remaley AT, Staels B, Stroes ESG, Taskinen MR, Tokgozoglu LS, Tybjaerg-Hansen A, Stock JK, Catapano AL. Triglyceride-rich lipoproteins and their remnants: metabolic insights, role in atherosclerotic cardiovascular disease, and emerging therapeutic strategies-a consensus statement from the European Atherosclerosis Society. Eur Heart J. 2021 Dec 14;42(47):4791-4806. doi: 10.1093/eurheartj/ehab551. PMID 34472586
- [Background] Mach F, Baigent C, Catapano AL, Koskinas KC, Casula M, Badimon L, Chapman MJ, De Backer GG, Delgado V, Ference BA, Graham IM, Halliday A, Landmesser U, Mihaylova B, Pedersen TR, Riccardi G, Richter DJ, Sabatine MS, Taskinen MR, Tokgozoglu L, Wiklund O; ESC Scientific Document Group. 2019 ESC/EAS Guidelines for the management of dyslipidaemias: lipid modification to reduce cardiovascular risk. Eur Heart J. 2020 Jan 1;41(1):111-188. doi: 10.1093/eurheartj/ehz455. No abstract available. PMID 31504418
- [Background] Grundy SM, Stone NJ, Bailey AL, Beam C, Birtcher KK, Blumenthal RS, Braun LT, de Ferranti S, Faiella-Tommasino J, Forman DE, Goldberg R, Heidenreich PA, Hlatky MA, Jones DW, Lloyd-Jones D, Lopez-Pajares N, Ndumele CE, Orringer CE, Peralta CA, Saseen JJ, Smith SC Jr, Sperling L, Virani SS, Yeboah J. 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Jun 18;139(25):e1082-e1143. doi: 10.1161/CIR.0000000000000625. Epub 2018 Nov 10. PMID 30586774
- [Background] Yannakoulia M, Scarmeas N. Diets. N Engl J Med. 2024 Jun 13;390(22):2098-2106. doi: 10.1056/NEJMra2211889. No abstract available. PMID 38865662
- [Background] Delgado-Lista J, Alcala-Diaz JF, Torres-Pena JD, Quintana-Navarro GM, Fuentes F, Garcia-Rios A, Ortiz-Morales AM, Gonzalez-Requero AI, Perez-Caballero AI, Yubero-Serrano EM, Rangel-Zuniga OA, Camargo A, Rodriguez-Cantalejo F, Lopez-Segura F, Badimon L, Ordovas JM, Perez-Jimenez F, Perez-Martinez P, Lopez-Miranda J; CORDIOPREV Investigators. Long-term secondary prevention of cardiovascular disease with a Mediterranean diet and a low-fat diet (CORDIOPREV): a randomised controlled trial. Lancet. 2022 May 14;399(10338):1876-1885. doi: 10.1016/S0140-6736(22)00122-2. Epub 2022 May 4. PMID 35525255